CLINICAL TRIAL: NCT00906854
Title: Urinary Incontinence and Practice of Physical Exercises Among Nulliparous and Nulligest Women
Brief Title: Urinary Incontinence and Practice of Physical Exercises
Status: Completed | Type: Observational
Sponsor: Universidade de Franca (Other)
Responsible Party: Lislei Jorge Patrizzi, Universidade de Franca
Other Study IDs: 0061/08
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; physical exercise
MeSH Terms: conditions — Urinary Incontinence; Motor Activity

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group I: practice of weight training exercises
- Group II: aerobic exercises as part of lessons jump, step and dance classes
- Group III: swimming (crawl mode)

SUMMARY:
Introduction: Urinary incontinence is often seen as a problem that affects multipara and old-aged women, however, there is evidence that during high impact physical activity, mainly, or those ones which promote a sudden increase of intra-abdominal pressure, this symptom is common, even among young women, physically active, and without known risk factors.

Objective: Evaluate the prevalence of urinary incontinence in nulliparous and nulligest women who regularly practice physical activities.

Method: 108 women, nulliparous and nulligest, average age 23.9 years old (from 18 to 30 years old) who exercise regularly. They were divided into 3 groups according to the regular practice of exercise forms, they are (G1) weight training, (G2) aerobic exercises, included jump, step and dancing classes, and (G3) swimming (crawl mode). All participants were questioned about the perception of leakage of urine during the practice of exercises. The established exclusion criterion included: surgeries of urinary tract, urinary infections, gestations, child-birth, advanced aged, obesity, sedentariness and practice of only one form of physical activity.

DETAILED DESCRIPTION:
The assessment was carried out in academies of the city of Franca. All participants were questioned about the perception of loss of urine during the practice of exercises.

ELIGIBILITY:
Inclusion Criteria:

* practice of exercises

Exclusion Criteria:

* surgeries of urinary tract
* urinary infections
* gestations
* child-birth
* advanced aged
* obesity
* sedentary and practice of only one form of physical activity

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 108 women, nulliparous and nulligest, average age 23.9 years old (from 18 to 30 years old) who exercise regularly. They were divided into 3 groups according to the regular practice of exercise forms, they are (G1) weight training, (G2) aerobic exercises, included jump, step and dancing classes, and (G3) swimming. All participants were questioned about the perception of leakage of urine during the practice of exercises.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lislei Patrizzi, Study Director — Universidade de Franca